CLINICAL TRIAL: NCT07155889
Title: Waste Management With Educational Competition Method in Nursing Students: A Randomized Controlled Trial
Brief Title: Educational Competition for Waste Management in Nursing Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SÜMEYYE BİLGİLİ TEKİN (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor-Investigator, SÜMEYYE BİLGİLİ TEKİN, Nursing Fundamentals Graduate Student, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AU-SBİLGİLİ_002
Record Dates: First submitted 2025-04-10; First posted 2025-09-04 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Waste Management
Keywords: Waste; Nursing; Nursing students; Teaching

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group using the educational competition method (Experimental): Pre-Test:
  Students are informed, consent is obtained, introductory information form and 'Knowledge Level Test' are applied.
  Training:
  Waste management training is given interactively by the researcher in 2 hours.
  Intervention (Educational Competition):
  A competition is organised with model wastes and colourful boxes.
  Students place the wastes in the correct boxes in 2 minutes.
  Observation, individual feedback and rewarding are made.
  Final Test and Satisfaction:
  After 1 week, 'Knowledge Level Test' and 'Satisfaction Form' are applied.
  Interventions: Other: Educational Competition Method
- Group Receiving Traditional Education (No Intervention): Pre-Test:
  Information, consent, introductory information form and 'Knowledge Level Test' are applied.
  Training:
  Waste management is explained by traditional method (no intervention).
  Post Test:
  After 1 week, only 'Knowledge Level Test' is applied.

INTERVENTIONS:
Other: Educational Competition Method — This study aims to evaluate nursing students' knowledge levels, practical skills, and the effectiveness of the educational competition method regarding medical waste management. The study consisted of three phases. In the first phase, students were informed, their consent was obtained, the "Informative Information Form" was completed, and the "Knowledge Level Test" was administered as a pre-test. In the second stage, the researcher gave a two-hour interactive lecture to all students, explaining the waste classification and separation processes. In the third stage, the "Educational Competition Method" was applied in Section A. In an arrangement prepared with mock waste and color-coded bins, students placed the waste in the appropriate bins within the specified time. The winner was rewarded at the end of the competition. One week later, a final test and satisfaction form were administered to evaluate the effectiveness of the method.
  Arms: Group using the educational competition method

SUMMARY:
The aim of this study is to investigate the effect of training nursing students on waste management through an educational competition method on their knowledge and satisfaction levels compared to the traditional method. During the training process, students will learn the correct classification of waste and reinforce this knowledge in a practical competition environment. The study is designed in a randomized controlled experimental design and experimental and control groups will be compared. Data collection tools will include "Student Introductory Information Form," "Knowledge Level Test" and "Student Satisfaction Evaluation Form." As a result of the study, it is expected that the educational competition method will increase the level of knowledge and satisfaction of nursing students about waste management compared to the traditional education method. This study aims to demonstrate the effectiveness of educational competition as an innovative method in educational approaches for nursing students.

DETAILED DESCRIPTION:
Type of Research: This research was designed as a randomized controlled pretest-posttest experimental study.

Location and Characteristics of the Research: There are three departments in the Faculty of Nursing at Atatürk University. There are 90 students in each department in the fourth year.

Research Population and Sample The research population consists of 270 students in the fourth year of the nursing department. As part of accreditation, each branch attends classes in the same classroom, and the same faculty member teaches the subject using the same method. To prevent contamination between the intervention and control groups, one group will be designated as the intervention group and one as the control group. To determine which group is the intervention group and which is the control group, the names of the three branches will be written on pieces of paper and drawn by lottery. The sample size was calculated using the GPower 3.1.9.2 program, with a margin of error of 0.05 and 80% test power, determining that at least 30 students per group would be sufficient. The research sample will consist of a total of 60 students, including 30 intervention and 30 control students who volunteer to participate in the research and meet the inclusion criteria. To account for possible data loss, 35+35=70 students will be recruited.

Research Inclusion Criteria

* Be over 18 years of age
* Being a 4th-year student
* Not having transferred horizontally or vertically
* Not having been absent during the dates when the research data will be collected Exclusion Criteria for the Research

  * Those who are not 4th-year nursing students
  * Students who have transferred horizontally/vertically
  * Students who graduated from a Health Vocational High School Data Collection Tools Data The "Student Identification Information Form," "Knowledge Level Test," and "Student Satisfaction Evaluation Form" will be used to collect data.

Student Identification Information Form (APPENDIX 1) This form was prepared by researchers in line with the literature and contains questions that inquire about the demographic characteristics of students, such as age, gender, socioeconomic level, etc.

Knowledge Level Test (Appendix 2) Multiple-choice questions will be prepared by researchers based on a literature review. A "Knowledge Level Test" covering the topic of waste management will be created. The Knowledge Level Test, consisting of 25 multiple-choice questions deemed appropriate for the purpose of the research, will be reproduced in quantities equal to the number of students and kept ready before the application.

Students participating in the research will be brought to the classroom and given the "Knowledge Level Test (pre-test)". Knowledge level tests will be evaluated on a scale of 100 points. The Knowledge Level Test results will be evaluated by awarding "4" points for each correct answer and "0" points for each incorrect answer. The highest score students can achieve on the achievement tests is '100' and the lowest score is "0".

The Knowledge Level Test will not be used as a performance grade/evaluation grade for students. The questions will be prepared specifically for this research for the first time. Furthermore, these prepared questions will not be used in the students' midterm/final exams. This information will also be disclosed to the students. The knowledge level tests will be reviewed by five faculty members specializing in the Department of Nursing Fundamentals. The questions submitted for expert review will be finalized after incorporating the necessary suggestions.

Student Satisfaction Evaluation Form (Appendix 3) This form, used to evaluate student satisfaction with the education program, was developed by the researchers through a literature review (Dilcen et al. 2023; Pourghaznein et al. 2015). This form has a 5-point Likert-type rating scale: (1) strongly disagree, (2) disagree, (3) undecided, (4) agree, and (5) strongly agree. To evaluate the form's clarity and functionality, five experts in the field of Nursing Fundamentals will be consulted to finalize the form.

Educational Competition Method The educational competition method will be used for waste management training to teach nursing students this skill, which is critical in patient care, in detail. In this training, students will gain knowledge and skills on the management of various wastes and how these wastes can be integrated into clinical decision-making processes.

Waste management training is structured using an educational competition method and aims to develop nursing students' knowledge and skills regarding the classification of medical waste. The training process will begin with theoretical instruction. Students will be provided with detailed information about the types of medical waste (biological waste, sharps waste, recyclable waste, and household waste), focusing on how these wastes should be classified and the risks that incorrect classification can pose. In addition, the color-coded waste bins designated for each type of waste and the procedures for using these bins will be explained. Following the theoretical briefing, a practical competition will be organized for the students.

The competition will be held in a setting featuring mock medical waste and waste bins. In the competition:

* Students will be taken to the setup in turn and asked to classify the waste correctly within a specified time.
* Each student will attempt to place the mock waste into the appropriately color-coded waste bins within the given time.
* Students will work in small groups to collaborate on the given medical waste and attempt to complete the correct classification as quickly as possible.
* This process will contribute to the development of students' teamwork and communication skills.

Throughout the competition, researchers will observe the process and take notes on the students' performance. Any mistakes made by each student or group will be recorded, and detailed feedback will be provided at the end of the competition. This feedback will help students recognize their shortcomings in the classification process and reinforce their learning. At the end of the competition, individual and group performances will be evaluated, and the participants with the highest achievements will be rewarded. Small symbolic prizes aim to increase student motivation.

This method aims to increase students' awareness and practical skills in medical waste management while also providing a fun and interactive learning environment.

Data Collection The research will be conducted between February 2025 and July 2025. The research data will be collected during the spring semester of the 2024-2025 academic year. The research will be completed between February 2025 and December 2025.

In the first stage, all students will be informed about the research and their consent will be obtained. Students who give their informed consent and agree to participate in the research will fill out a "Student Identification Form" under observation in the classroom. Then, all students will take a "Knowledge Level Test" as a pre-test. It was determined that students took two hours of theoretical classes on public health in the nursing principles course and two hours on waste management over four years.

In the second stage, the topic of waste management will be presented interactively to all students by the same researcher for two hours per week.

Intervention Group (Section A) In the third stage, the educational competition method previously developed for this research will be used. The content of this educational competition method was developed by the researchers.

Educational Competition Method Objective: This educational competition method aims to increase nursing students' knowledge and practical skills in medical waste management, ensure they learn the correct waste separation processes, and reinforce what they have learned.

Materials and Equipment

* Model Waste: Various materials (e.g., bloody gauze, used needles, plastic bottles, gloves, etc.) representing all types of medical waste used in hospitals will be prepared as models. Each model will be designed and labeled to correspond to its real-life counterpart.
* Waste Bins: The setup will include color-coded waste bins with explanatory labels for biological waste, sharps waste, recyclable waste, and household waste.

Process Flow

1. Pre-Competition Briefing:

   * Students will be provided with theoretical information on the classification of medical waste, and each waste category will be explained in detail.
   * Students will be informed of the competition rules.
2. Implementation of the Competition:

   * Students will take turns at the station.
   * Each student will be given a specific amount of time (2 minutes). During this time, students will place the mock waste into the appropriate waste bins.
   * During the competition, researchers will observe the students' classification and take notes.
3. Evaluation and Feedback:

   * At the end of the competition, the students' rate of placing waste into the correct bins will be evaluated.
   * Researchers will provide detailed feedback by individually analyzing the students' correct and incorrect actions during the classification process. This feedback process will create a structured learning environment for students to recognize their mistakes and improve their learning.
4. Rewards:

   * Students who classify the most correctly will be encouraged with a small reward. This reward aims to increase motivation in the competition environment.

One week after the competition, the "Knowledge Level Test" will be administered as the final test, and student satisfaction will be assessed using the "Student Satisfaction Evaluation Form." Control Group (Section C) In the fourth stage, No intervention will be made. The topic of waste management will be explained using traditional methods.

In the fifth stage, the "Knowledge Level Test" will be administered as the final test to students in both the intervention and control groups one week after the training.

Data Evaluation The SPSS 23.0 (Statistical Programme for Social Sciences) package program will be used to evaluate the data obtained from the research. The normality of the variables will be examined using visual (histograms, probability plots) and analytical methods (Kolmogorov-Smirnov test). When comparing the control and intervention groups, the independent groups t-test will be used for comparisons between continuously distributed variables that show a normal distribution, and the chi-square test will be used for categorical variables. If the data from the comparison of the scale scores before and after the intervention in the intervention group show a normal distribution, the paired t-test will be applied; if they do not show a normal distribution, the Wilcoxon test will be applied. The relationships between variables will be evaluated using Pearson correlation analysis for values showing a normal distribution and Spearman correlation analysis for those not showing a normal distribution. The statistical significance level will be accepted as p<0.05.

The evaluation of the results and the statistical analyses are the responsibility of the research supervisor and the research team. Statistics will be evaluated using the blinding method. Data will be collected by the researcher. In order not to jeopardize the reliability of the research at the data analysis stage, data will be obtained from a professional company. Entering the data collected by the researcher into the SPSS system and performing the analysis will be carried out by obtaining services from professional companies. The accuracy of the analyses will be evaluated by statistics experts before and after the analyses are performed, and the results will be evaluated with other faculty members who are experts in the field.

Difficulties and Limitations of the Research:

The fact that this research is conducted only with 4th-year nursing students studying at a university nursing faculty constitutes a limitation of the research. Furthermore, the possibility of interaction between students in the intervention and control groups increases the limitations of the research.

Ethical Principles of the Research Before starting the research, approval will be obtained from the Ethics Committee of Atatürk University Faculty of Nursing. After obtaining the ethics committee approval, institutional permission will be obtained from Atatürk University Faculty of Nursing. During the collection of research data, written and verbal consent will be obtained by informing individuals about the research in accordance with the principle of "Informed Consent," stating that they are free to participate or not participate in the research in accordance with the principle of "Respect for Autonomy," and stating that the information of individuals participating in the research will be kept confidential in accordance with the principle of "Confidentiality and Protection of Confidentiality." Those willing to participate in the research will be included in the scope of the research. Since individual rights must be protected in the research, the Helsinki Declaration on Human Rights will be adhered to during the study period.

It will be stated that the research results will not affect any performance evaluation, midterm and final grades, and that the educational competition method will be applied to the control group in the same way after the research is completed.

Variables of the Study Dependent Variables Knowledge Level Tests are the dependent variables of the study. Independent Variables The application of the Educational Competition Method is the independent variable of the study.

ELIGIBILITY:
Inclusion Criteria

* Being over 18 years of age
* Being a 4th year student
* Not being a horizontal or vertical transfer student
* Not being absent on the dates when the research data will be collected Exclusion Criteria
* Not being a 4th year nursing student
* Students who come with horizontal/vertical transfer
* Students graduating from Health Vocational High School

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-11-10 (Estimated)

PRIMARY OUTCOMES:
Student Information Form | 2 weeks
  This form has been prepared by researchers in accordance with the literature and contains questions that inquire about the demographic characteristics of students, such as age, gender, socioeconomic status, etc.
Knowledge Level Test | 2 weeks
  Multiple-choice questions will be prepared by researchers based on a literature review. A Knowledge Level Test will be created on the subject of waste management. The Knowledge Level Test, consisting of 25 multiple-choice questions deemed appropriate for the purpose of the research, will be reproduced in quantities equal to the number of students and kept ready before the application.
  Students participating in the research will be brought into the classroom, and the "Knowledge Level Test (pre-test)" will be administered. The evaluation of the knowledge level tests will be conducted on a scale of 100 points. The Knowledge Level Test results will be evaluated by awarding "4" points for each correct answer and '0' points for each incorrect answer. The highest possible score students can achieve on the achievement tests is "100," and the lowest possible score is "0."
Student Satisfaction Evaluation Form | 2 weeks
  This form, used to evaluate student satisfaction with the education program, was developed by researchers through a literature review. The form has a 5-point Likert-type scale with the following options: (1) strongly disagree, (2) disagree, (3) undecided, (4) agree, and (5) strongly agree. The final version of the form will be determined after obtaining opinions from five experts in the field of Nursing Fundamentals to evaluate its clarity and functionality.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No